CLINICAL TRIAL: NCT07134959
Title: Validity and Reliability of Turkish Version Exercise Benefits/Barriers Scale in Pregnant Women
Brief Title: Exercise Benefits and Barriers in Pregnancy
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Semiha Yenişehir, Principal Investigator, Ordu University
Other Study IDs: E-1146814
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy
Keywords: pregnancy; exercise; Questionnaire; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: pregnant women
- control group: healthy non-pregnant women

SUMMARY:
The aim of this study is to examine the validity and reliability of the Exercise Benefits/Barriers Scale in pregnant women. It will contribute to raising awareness about engaging in physical activity and exercise during pregnancy in the pregnant population through the applied questionnaires.

DETAILED DESCRIPTION:
Regular physical activity (PA) and exercise during pregnancy help protect the health of both the mother and the baby by reducing the risk of excessive gestational weight gain, hypertension, gestational diabetes, venous problems, and birth-related complications. They also have positive effects on sleep, stress, anxiety, depression, and overall quality of life. However, PA participation rates during pregnancy are low and tend to decline as pregnancy progresses through the trimesters. Hormonal and physiological changes, weight gain, fatigue, and psychological disturbances are among the main factors limiting participation. Therefore, identifying the barriers to PA during pregnancy and developing strategies to address them is essential. Assessing perceptions of the benefits and barriers to exercise can guide interventions aimed at increasing PA levels. This study aims to determine the validity and reliability of the Exercise Benefits/Barriers Scale in pregnant women, with the expectation that its findings will provide valuable evidence for both scientific research and clinical practice.

ELIGIBILITY:
Inclusion Criteria for Study Group:

1. Being between 18 and 45 years of age,
2. Being in the second or third trimester of pregnancy,
3. Being literate in Turkish,
4. Willingness to participate in the study.

Exclusion Criteria for Study Group:

1. Presence of pregnancy complications that may prevent physical activity and exercise (e.g., preeclampsia, vaginal bleeding, heart disease),
2. Presence of orthopedic or neurological problems that may hinder participation in the study,
3. Presence of visual, auditory, or cognitive impairments severe enough to prevent participation in the study,
4. Multiple pregnancy.

Inclusion Criteria for Control Group:

1. Being between 18 and 45 years of age,
2. Female sex,
3. Being literate in Turkish,
4. Willingness to participate in the study.

Exclusion Criteria for Control Group:

1. Having a disease severe enough to prevent physical activity and exercise (e.g., endocrine and metabolic disorders, cardiopulmonary diseases),
2. Presence of orthopedic or neurological problems that may hinder participation in the study,
3. Presence of visual, auditory, or cognitive impairments severe enough to prevent participation in the study,
4. Participation in another experimental or drug study during the study period,
5. Being pregnant or suspected of pregnancy,
6. Having experienced pregnancy, childbirth, or surgical intervention within the last six months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Study Population: Ordu University Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Exercise Benefits/Barriers Scale (EBBS): | At baseline and 5 days after the first assessment
  Developed in 1987 by Sechrist et al. to assess individuals' perceptions of the benefits of and barriers to exercise (Sechrist et al., 1987). It is a Likert-type scale with responses rated from "4 = strongly agree" to "1 = strongly disagree." The scale consists of two subscales: EBBS-Benefits and EBBS-Barriers. The EBBS-Benefits subscale contains 29 items, while the EBBS-Barriers subscale contains 14 items. In the EBBS-Barriers subscale, lower scores indicate a higher perceived barrier to exercise, whereas in the EBBS-Benefits subscale, higher scores indicate a more positive perception of exercise. The validity and reliability of the Turkish version were demonstrated by Saraç et al. (2024), with Cronbach's alpha coefficients of 0.95 for the EBBS-Benefits subscale and 0.82 for the EBBS-Barriers subscale (Saraç et al., 2024).

SECONDARY OUTCOMES:
Barriers to Physical Activity During Pregnancy Scale | at baseline
  Developed by Amiri-Farahani et al. (2021) to evaluate barriers to physical activity among pregnant women. The scale consists of 29 items and four subdimensions, with each item scored on a 5-point Likert scale (1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree). Higher scores indicate greater barriers to physical activity (Amiri-Farahani et al., 2021). The validity and reliability of the Turkish version were confirmed by Ataman Bor and Hanligil, with Cronbach's alpha coefficients reported as follows: total scale, 0.91; pregnancy-related personal barriers, 0.88; non-pregnancy-related personal barriers, 0.89; interpersonal barriers, 0.87; environmental barriers, 0.80 (Bor & Hanligil, 2024).
Pregnancy Physical Activity Questionnaire (PPAQ) | at baseline
  Developed by Chasan-Taber et al. (2004), this semi-quantitative questionnaire asks participants to report the amount of time spent on 32 different activities. These include household/caregiving activities (13 items), occupational activities (5 items), sports/exercise (8 items), transportation (3 items), and inactivity (3 items). For each activity, participants indicate the amount of time they typically spend per day or week during their current trimester. Time intervals range from 0 to 6 or more hours per day and 0 to 3 or more hours per week. An open-ended section at the end allows participants to list other activities not included in the questionnaire. Weekly total energy expenditure is calculated as MET-hours/week (Chasan-Taber et al., 2004). The Turkish validity and reliability study was conducted by Çırak et al. (2015).
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | at baseline
  Physical activity levels will be assessed using the Turkish version of the IPAQ-SF, which has demonstrated validity and reliability (Saglam et al., 2010). The questionnaire consists of seven items evaluating time spent in walking, moderate-intensity, and vigorous-intensity activities, as well as one separate question assessing time spent sitting. Scoring involves calculating total minutes and days for walking, moderate, and vigorous activities. MET-minutes are computed by multiplying the minutes spent in each activity by its MET value (vigorous activity = 8 METs, moderate activity = 4 METs, walking = 3.3 METs). Participants are classified into three categories based on total MET-minutes: "inactive," "minimally active," and "highly active" (Saglam et al., 2010).
Pregnancy Exercise Self-Efficacy Questionnaire | at baseline
  This 10-item questionnaire assesses pregnant women's perceived ability and motivation to engage in physical activity under various circumstances. Adapted from the Exercise Self-Efficacy Scale, it was developed by Brand et al. to explain and predict changes in exercise behavior. A 5-point Likert scale is used (1 = strongly disagree to 5 = strongly agree), with total scores ranging from 10 to 50. Scores are categorized as follows: low self-efficacy, 10-17 points; moderate self-efficacy, 18-34 points; high self-efficacy, 35-50 points (Brand et al., 2013). The Turkish validity and reliability study was conducted by Üzelpasaci et al. (2023), with a Cronbach's alpha of 0.889.
Visual Analog Scale (VAS) for Kinesiophobia | at baseline
  The severity of kinesiophobia among pregnant participants will be assessed using a vertical 0-10 cm Visual Analog Scale through the following question:
  • "I am afraid that exercising during pregnancy might harm my baby" (0 = not afraid at all, 10 = extremely afraid)
  Participants will be asked to mark a point on the VAS, and the distance from 0 will be measured with a ruler.

CONTACTS AND LOCATIONS:
Overall Officials: Semiha Yenişehir, Principal Investigator — Ordu University
Locations (1):
- Ordu Üniversitesi, Ordu, Altınordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No